CLINICAL TRIAL: NCT01529567
Title: Cognitive Behavioral Therapy With Our Without Exposure Therapy for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS-0
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT without exposure (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy without exposure
- CBT with exposure (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy with exposure

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy without exposure — 10 week internet-delivered cognitive behavioral therapy, including mindfulness training, education about the negative effects of excessive avoidance and control behaviors on IBS symptoms and quality of life, and guided behavioral change aiming to increase quality of life and flexibility.
  Arms: CBT without exposure
Behavioral: Cognitive Behavioral Therapy with exposure — 10 week internet-delivered cognitive behavioral therapy, including mindfulness training, education about the negative effects of excessive avoidance and control behaviors on IBS symptoms and quality of life, guided behavioral change aiming to increase quality of life and flexibility, and systematic exposure to IBS symptoms and aversive situations.
  Arms: CBT with exposure

SUMMARY:
Patients with a diagnosis of irritable bowel syndrome (IBS) are recruited by self-referral. They are randomized to two 10 weeks of internet-delivered cognitive behavioral programs. Both programs include mindfulness training, education about how excessive avoidant and control behaviors maintain IBS symptoms, and changing of these behaviors to live a richer life. One of the programs also includes instructions on how to perform systematic exposure. The hypothesis of the study is while both groups will show improvement in terms of IBS symptom severity and quality of life, the addition of systematic exposure will lead to more improvement in symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Fluency in Swedish
* IBS-diagnosis established by physician
* Fulfillment of Rome III criteria for IBS

Exclusion Criteria:

* Diarrhea predominance with no colonoscopy performed
* Blood in stool without benign medical explanation
* Rapid weight loss without benign medical explanation
* Ongoing alcohol or drug abuse
* Suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptom rating scale | 1 week before randomization
Gastrointestinal symptom rating scale | 10 weeks after randomization (i.e. after conclusion of treatment)
Gastrointestinal symptom rating scale | 36 weeks after randomization (i.e. 6 months after conclusion of treatment)

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Quality of Life Instrument (IBS-QOL) | 1 week before randomization
Irritable Bowel Syndrome Quality of Life Instrument (IBS-QOL) | 10 weeks after randomization (i.e. after conclusion of treatment)
Irritable Bowel Syndrome Quality of Life Instrument (IBS-QOL) | 36 weeks after randomization (i.e. 6 months after conclusion of treatment)
Visceral Sensitivity Index (VSI) | 1 week before randomization
Visceral Sensitivity Index (VSI) | 10 weeks after randomization (i.e. after conclusion of treatment)
Visceral Sensitivity Index (VSI) | 36 weeks after randomization (i.e. 6 months after conclusion of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, PhD, Principal Investigator — Karolinska Institutet

REFERENCES:
- [Derived] Wallen H, Lindfors P, Andersson E, Hedman-Lagerlof E, Hesser H, Lindefors N, Svanborg C, Ljotsson B. Return on investment of internet delivered exposure therapy for irritable bowel syndrome: a randomized controlled trial. BMC Gastroenterol. 2021 Jul 13;21(1):289. doi: 10.1186/s12876-021-01867-6. PMID 34256715